CLINICAL TRIAL: NCT02318888
Title: Does Icodextrin Reduce the Risk of Small Bowel Obstruction?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 2009/123
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Surgical Adhesions
Keywords: Small bowel obstruction, Surgery, Colorectal cancer
MeSH Terms: conditions — Tissue Adhesions; Colorectal Neoplasms | interventions — Surgical Procedures, Operative; Icodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery and Icodextrin (Experimental): Icodextrin 4% instilled every 30 minutes during surgery and 1000 ml instilled before closure of abdomen
  Interventions: Procedure: Surgery; Drug: Icodextrin
- Surgery (Active Comparator): No instillations during surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery
Drug: Icodextrin
  Arms: Surgery and Icodextrin

SUMMARY:
The study aims at investigating if icodextrin 4% instilled in abdominal cavity during surgery can reduce the risk of surgery and hospitalisation for small bowel obstruction in patients with colorectal cancer. Follow-up data is collected from the Swedish national colorectal cancer registry.Patients are followed for 5 years postoperatively.The study is a randomized Swedish multicenter study and planned to include 1,800 patients. A safety control is planned after 300 included patients.

DETAILED DESCRIPTION:
Icodextrin 7.5% is used in peritoneal dialysis. In animal models and in gynecological surgery a 4% solution of Icodextrin has been tested as a possible agent of reducing adhesions by acting as a barrier between peritoneal surfaces. Some data support a reduction af adhesions (van den Tool et al., Brown et al.). However, is not known whether icodextrin reduces the need for surgery or hospitalisation for small bowel obstruction.This study aims to study these parameters as well as complications and survival.

Patients with colorectal cancer and scheduled for surgery with curative intent will be (after patients acceptance) randomized to have icodextrin 4% instilled in the abdominal cavity or not. Patients allocated to icodextrin arm will have 100 ml of icodextrin 4% instilled every 30 minutes during surgery and at end of operation further 1000 ml instilled in the abdominal cavity. Postoperative care is performed according to each hospital praxis.

Follow-up data will be collected from the Swedish National Colorectal cancer registry. Data 30 days postoperatively will be analysed for early small bowel obstruction and other early complications. The study ends 5 years postoperatively with analysis of surgery and hospitalization for small bowel obstruction as well as survival and longterm complications.

A safety analysis is planned after the first 300 randomized patients with respect to early (30 days) complications. These data will analysed blindly by external reviewers.

Randomization (1:1) will be performed at the Regional Cancer Centrum in the Uppsala-Örebro region. The study aims to randomise 1800 patients.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer
* Curative surgery planned
* Informed consent
* Age 18-85

Exclusion Criteria:

* Local surgery planned
* Generalized disease
* Other malignancy
* Not informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1808 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Surgery for small bowel obstruction | 5 years
  The proportion of patients that have undergone surgery for small bowel obstruction will be compared between the groups.

SECONDARY OUTCOMES:
Hospitalisation for small bowel obstruction | 5 years
Overall and cancer survival | 5 years
Postoperative complications | 30 days
  Safety control of first 300 randomised patients
Postoperative complications | 30 days
  For all randomised patients

CONTACTS AND LOCATIONS:
Overall Officials: Urban Karlbom, PhD, Principal Investigator — University Hospital, Uppsala; Lars Påhlman, Professor, Study Director — University Hospital
Locations (13):
- Sweden (13):
  - Eskilstuna Hospital, Eskilstuna
  - Falun Hospital, Falun
  - Gävle Hospital, Gävle
  - Jönköping Hospital, Jönköping
  - Karlstad Hospital, Karlstad
  - Lidköping Hospital, Lidköping
  - Luleå Hospital, Luleå
  - Mora Hospital, Mora
  - Norrrköping Hospital, Norrköping
  - Nyköping Hospital, Nyköping
  - Torsby Hospital, Torsby
  - University Hospital, Uppsala
  - Västerås Hospital, Västerås

REFERENCES:
- [Background] van den Tol P, ten Raa S, van Grevenstein H, Marquet R, van Eijck C, Jeekel H. Icodextrin reduces postoperative adhesion formation in rats without affecting peritoneal metastasis. Surgery. 2005 Mar;137(3):348-54. doi: 10.1016/j.surg.2004.06.001. PMID 15746791
- [Background] Brown CB, Luciano AA, Martin D, Peers E, Scrimgeour A, diZerega GS; Adept Adhesion Reduction Study Group. Adept (icodextrin 4% solution) reduces adhesions after laparoscopic surgery for adhesiolysis: a double-blind, randomized, controlled study. Fertil Steril. 2007 Nov;88(5):1413-26. doi: 10.1016/j.fertnstert.2006.12.084. Epub 2007 Mar 26. PMID 17383643
- [Derived] Sakari T, Sjodahl R, Pahlman L, Karlbom U. Role of icodextrin in the prevention of small bowel obstruction. Safety randomized patients control of the first 300 in the ADEPT trial. Colorectal Dis. 2016 Mar;18(3):295-300. doi: 10.1111/codi.13095. PMID 26934850